CLINICAL TRIAL: NCT03427762
Title: Compare the Effects of Agility and Cycling Exercise Training on Mobility and Balance in PD and Healthy Old Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Principal Investigator, Tollár József, Principal Investigator, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKEB009/2017
Record Dates: First submitted 2018-02-03; First posted 2018-02-09 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2018-02

CONDITIONS: Healthy; Movement Disorders; Parkinson Disease; Condition
Keywords: balance; postural controll; motor controll; posturgraphy; quality of life
MeSH Terms: conditions — Movement Disorders; Parkinson Disease; Disease | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy cycling group (Experimental): During a 5-week intervention, we examine the patients' balance, postural control, quality of life and mobility. Then there is a bicycle every 1 hour.
  Interventions: Other: Rehabilitation
- Healthy xbox group (Experimental): During a 5-week intervention, we examine the patients' balance, postural control, quality of life and mobility. Then they will train 1 hour every day on an xbox program.
  Interventions: Other: Rehabilitation
- Healthy controll group (No Intervention): During a 5-week intervention, we examine the patients' balance, postural control, quality of life and mobility. Thereafter, the group does not move only in everyday life.
- PD groupe (Experimental): Patients with PD have already been evaluated and compared to the results of a healthy group within a separate experiment.
  The study and the results have been completed. Clinical trial number:NCT03193268
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Healthy cycling group: The group participates in 5 weeks of intensive cycling therapy.
  Healthy xbox group: The group participates in 5 week intensive xbox therapy Healthy controll group: The group does not take any kind of therapy. PD group: We have already analyzed the results of our group, and we will compare their results with the results of healthy groups.
  Other Names: Healthy cycling group; Healthy xbox group; PD group
  Arms: Healthy cycling group; Healthy xbox group; PD groupe

SUMMARY:
The purpose of the study is to compare the effectiveness and specificity of agility and cycling exercise training on balance and mobility outcomes in PD and age and gender matched healthy controls. The hypothesis is that due to being profoundly deconditioned, agility and cycling will be similarly effective in PD but agility will be more effective then cycling in healthy old adults, in improving mobility and balance.

ELIGIBILITY:
Inclusion Criteria:

* family doctor should be qualified as healthy.
* older adults had to have basic fitness
* weekly movement of at least 3 hours

Exclusion Criteria:

* Severe heart problems
* severe demeanor
* alcoholism
* drug problems

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-02-03 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Postural instability | 5 weeks
  Body sway (mm) (Posturography test)
quality of life | 5 weeks
  EQ-5D (EQ-5D was first introduced in 1990 by the EuroQol Group, The EQ-5D questionnaire is made up for two components; health state description and evaluation)
balance test | 5 weeks
  Berg Balance test (The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks, 41-56 = low fall risk, 21-40 = medium fall risk, 0 -20 = high fall risk )
mobility test | 5 weeks
  Six minutes walk test (6MWT) (m) (The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway)

SECONDARY OUTCOMES:
depression scale | 5 weeks
  Beck Depression scale (The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression, 0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, 29-63: severe depression)

CONTACTS AND LOCATIONS:
Overall Officials: József Tollár, MSC, Principal Investigator — Somogy Megyei Kaposi Mór Teaching Hospital
Locations (1):
- József Tollár, Kaposvár, Somogy County, Hungary

REFERENCES:
- [Derived] Tollar J, Nagy F, Moizs M, Toth BE, Sanders LMJ, Hortobagyi T. Diverse Exercises Similarly Reduce Older Adults' Mobility Limitations. Med Sci Sports Exerc. 2019 Sep;51(9):1809-1816. doi: 10.1249/MSS.0000000000002001. PMID 30973482
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=healthy+adult+training